CLINICAL TRIAL: NCT00413361
Title: Study of the Reduction of Systemic Lupus Erythematosus Flares Through Adaptation of the Dosage of Hydroxychloroquine to Its Whole-blood Concentration. National Multicenter Randomized Prospective Study
Brief Title: The Reduction of Systemic Lupus Erythematosus Flares :Study PLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Zakia IDIR, Department Clinical Rechearch of Developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P051070
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2007-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Hydroxychloroquine
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): placebo
  Interventions: Drug: versus hydroxychloroquine
- B (Experimental): versus hydroxychloroquine
  Interventions: Drug: versus hydroxychloroquine

INTERVENTIONS:
Drug: versus hydroxychloroquine — versus hydroxychloroquine

SUMMARY:
The main objective of study PLUS is to determine the potential benefits of individualized HCQ dosing schedules aimed at maintaining the whole-blood HCQ concentration above 1000 ng/ml

DETAILED DESCRIPTION:
Hydroxychloroquine (HCQ) is a treatment which allows preventing Systemic Lupus Erythematosus (SLE) exacerbations.

HCQ can be measured in whole-blood by HPLC (High Performance Liquid Chromatography).

Interindividual variability in blood HCQ concentrations is important and a correlation between HCQ level and clinical efficacy of HCQ has been demonstrated in SLE in a monocentric study of 143 unselected SLE patients.

The main objective of study PLUS is to determine the potential benefits of individualized HCQ dosing schedules aimed at maintaining the whole-blood HCQ concentration above 1000 ng/ml

The secondary objectives are:

* To define biological and clinical hallmarks present at M1 (month 1) which are predictor of SLE exacerbations in the next 6 month,
* To establish the parameters of HCQ pharmacokinetic model, by a study of population, using a "Bayésienne" approach.
* To study the influence of allelic variants of drug carriers and other genes in the interindividual variability of blood HCQ concentrations.
* To study the influence of the compliance in the blood HCQ concentration variability
* To study the relation between blood HCQ concentrations, SLE activity and quality of life
* To study the relation between blood HCQ concentrations, SLE activity and lipid profile of the patients
* To study the relation between ECG abnormalities and blood HCQ concentrations
* To constitute a bank of serum, a DNAbank, and a RNAbank to permit subsequent studies

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and above
* Diagnosis of Systemic Lupus Erythematosus (SLE) according to the American College of Rheumatology (ACR) Classification Criteria.
* Treatment with HCQ for at least 6 months, without modification of HCQ dosage for 2 months
* Stable dosage of HCQ from one day to another (200 g x 2/day or 400 mg once a day or 200 mg once a day)
* No increase in the steroids dosage during the 3 previous weeks
* Steroids dosage lower or equal to 0. 5 mg/kg/day of prednisone equivalent
* No modifications of a possible immunosuppressor during the 2 previous months
* SELENA-SLEDAI < or = 12
* Signature of the consent of participation

Exclusion Criteria:

* Known retinopathy, present or passed
* Severe cataract obstructing the ophthalmologic monitoring
* MONOPHTALM patients
* Past history of intolerance with HCQ (in particular gastro-intestinal, or retinal) during the possible former use of a higher dosage
* Use of nivaquine during the 3 previous months
* Treatment with biotherapy (for example Rituximab) during the 12 previous months
* Calculated clearance of creatinin lower than 60 ml/min
* Chronic alcoholism
* Liver failure
* Desire of pregnancy in the next 7 months
* Known non compliance, and risks of random follow-up
* Absence of social security cover

People profiting from a particular protection:

* Pregnant women
* Age under 18
* Patient under supervision and TRUSTEESHIP
* People who are hospitalized without their consent and not protected by the law
* People who are private of freedom.

Criteria of inclusion at the visit of randomization (D0):

All the patients responding to the next criterions can be randomized:

* Blood HCQ concentration ranging between 100 and 750 ng/ml at the time of the visit of preselection,
* No increase in the steroids dosage since last visit
* No modifications of a possible immunosuppressor since last visit
* SELENA-SLEDAI < or = 12 Activity of the lupus remaining stable (no increase of more than 2 points of the SELENA-SLEDAI),
* Ophthalmologic examination in the 6 previous months with no contra-indication for the use of HCQ,
* Absences of conductive disorders on the ECG
* Use of an effective contraception,
* Negative Beta-HCG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The number of patient in each group who developed a flare (according to the SELENA-SLEDAI composite criteria) during the study period. | 7 months of follow up
  The number of patient in each group who developed a flare (according to the SELENA-SLEDAI composite criteria) during the study period.

SECONDARY OUTCOMES:
The number of patients in each group who developed a flare during the study period. | 7 months of follow up
  The number of patients in each group who developed a flare during the study period.
The total number of flares in each group | 7 months of follow up
  The total number of flares in each group
the total dose of steroids in each group | 7 months of follow up
  the total dose of steroids in each group
the area under the curve of SELENA SLEDAI in each group | 7 months of follow up
  the area under the curve of SELENA SLEDAI in each group
the mean change of the quality of life questionnaire SF-36 | 7 months of follow up
  the mean change of the quality of life questionnaire SF-36
the mean change on the score of analogical visual scale in each group | 7 months of follow up
  the mean change on the score of analogical visual scale in each group
Treatment tolerance evaluation will include clinical, electrocardiographic and ophthalmologic screening. | 7 months of follow up
  Treatment tolerance evaluation will include clinical, electrocardiographic and ophthalmologic screening.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie COSTEDOAT-CHALUMEAU, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Chu Pitie Salpetriere, Paris
  - Hopital la Pitié Salpétrière Assistance Publique, Paris

REFERENCES:
- [Derived] Morris DL, Sheng Y, Zhang Y, Wang YF, Zhu Z, Tombleson P, Chen L, Cunninghame Graham DS, Bentham J, Roberts AL, Chen R, Zuo X, Wang T, Wen L, Yang C, Liu L, Yang L, Li F, Huang Y, Yin X, Yang S, Ronnblom L, Furnrohr BG, Voll RE, Schett G, Costedoat-Chalumeau N, Gaffney PM, Lau YL, Zhang X, Yang W, Cui Y, Vyse TJ. Genome-wide association meta-analysis in Chinese and European individuals identifies ten new loci associated with systemic lupus erythematosus. Nat Genet. 2016 Aug;48(8):940-946. doi: 10.1038/ng.3603. Epub 2016 Jul 11. PMID 27399966
- [Derived] Schoindre Y, Jallouli M, Tanguy ML, Ghillani P, Galicier L, Aumaitre O, Frances C, Le Guern V, Liote F, Smail A, Limal N, Perard L, Desmurs-Clavel H, Le Thi Huong D, Asli B, Kahn JE, Sailler L, Ackermann F, Papo T, Sacre K, Fain O, Stirnemann J, Cacoub P, Leroux G, Cohen-Bittan J, Hulot JS, Lechat P, Musset L, Piette JC, Amoura Z, Souberbielle JC, Costedoat-Chalumeau N; Group PLUS. Lower vitamin D levels are associated with higher systemic lupus erythematosus activity, but not predictive of disease flare-up. Lupus Sci Med. 2014 Jun 7;1(1):e000027. doi: 10.1136/lupus-2014-000027. eCollection 2014. PMID 25379192
- [Derived] Morel N, Bachelot A, Chakhtoura Z, Ghillani-Dalbin P, Amoura Z, Galicier L, Aumaitre O, Piette JC, Pourrat J, Boutin D, Sacre K, Kahn JE, Duhaut P, Farge D, Frances C, Guettrot-Imbert G, Harle JR, Lambotte O, Le Guern V, Sene D, Trad S, Vidal E, Sarrot-Reynauld F, Gompel A, Tanguy ML, Touraine P, Lacorte JM, Costedoat-Chalumeau N; PLUS group. Study of anti-Mullerian hormone and its relation to the subsequent probability of pregnancy in 112 patients with systemic lupus erythematosus, exposed or not to cyclophosphamide. J Clin Endocrinol Metab. 2013 Sep;98(9):3785-92. doi: 10.1210/jc.2013-1235. Epub 2013 Jul 5. PMID 23833039
- [Derived] Costedoat-Chalumeau N, Galicier L, Aumaitre O, Frances C, Le Guern V, Liote F, Smail A, Limal N, Perard L, Desmurs-Clavel H, Boutin du LT, Asli B, Kahn JE, Pourrat J, Sailler L, Ackermann F, Papo T, Sacre K, Fain O, Stirnemann J, Cacoub P, Jallouli M, Leroux G, Cohen-Bittan J, Tanguy ML, Hulot JS, Lechat P, Musset L, Amoura Z, Piette JC; Group PLUS. Hydroxychloroquine in systemic lupus erythematosus: results of a French multicentre controlled trial (PLUS Study). Ann Rheum Dis. 2013 Nov;72(11):1786-92. doi: 10.1136/annrheumdis-2012-202322. Epub 2012 Nov 10. PMID 23144449